CLINICAL TRIAL: NCT05339542
Title: Musculoskeletal Ultrasound Changes in the Plantar Fascia After a Single Injection of Platelet Rich Plasma Compared to Steroid
Brief Title: Platelet Rich Plasma in Plantar Fasciitis
Acronym: PRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahmed ElSayed Hafez, Principal investigator, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rheumatology Dep.
Record Dates: First submitted 2022-04-09; First posted 2022-04-21 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Plantar Fascitis
Keywords: degenerative plantar fasciitis; platelet rich plasma; ultrasound guided injection; heel pain; interventional rheumatology
MeSH Terms: interventions — Methylprednisolone

STUDY DESIGN:
Intervention Model Description: the study will include two groups. Group I (study group) will be injected PRP. Group II (control group) will be injected methylprednisolone
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelet rich plasma group (Experimental): platelet rich plasma (PRP) will be produced through whole blood centrifuge using a specific methodology in a strict aseptic setting. Then, blood will be collected and mixed with anticoagulant and Citrate-phosphate-dextrose adenine in a 10 volume blood to 1 volume anticoagulant ratio. The blood will be centrifuged for 10 minutes at 1000 rpm. Afterward, the plasma will be transferred to a new glass tube and centrifuged for 15 minutes at 3000 rpm. At the bottom of the tube, platelets will form a pellet. Finally, pure platelet-rich plasma will be obtained at a concentration of up to four times higher than baseline. Prior to the injection, calcium gluconate will be combined with PRP (at a ratio of 0.3 ml ca gluconate/ml PRP).
  The injection will be done once.
  Interventions: Other: platelet rich plasma
- Methylprednisolone group (Active Comparator): 2 ml methylprednisolone acetate 40mg/ml (total 80mg methylprednisolone acetate) together with 1 ml lidocaine 2% (total 3 ml solution) will be directly injected under ultrasound guidance to the plantar fascia.This group serves as active comparative group.
  The injection will be done once.
  Interventions: Drug: MethylPREDNISolone 40 MG

INTERVENTIONS:
Other: platelet rich plasma — derived from patient own blood
  Arms: Platelet rich plasma group
Drug: MethylPREDNISolone 40 MG — active comparative intervention
  Other Names: 1 ml Lidocaine 2%
  Arms: Methylprednisolone group

SUMMARY:
a number of patient diagnosed as degenerative plantar fasciitis will be collected and divided into two groups, group I will be injected by platelet rich plasma and group II will be injected methylprednisolone

DETAILED DESCRIPTION:
the study will include 100 patients diagnosed as degenerative plantar fasciitis and will be evaluated by musculoskeletal ultrasound by two observes and the will divided randomly into two groups who will be injected under ultrasound imaging by either Platelet rich plasma or methylprednisolone. selection of patient will be randomly and the study will be double blinded.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of plantar fasciitis

Exclusion Criteria (history or current):

* Rheumatic diseases
* Foot Trauma
* Neurological diseases
* Thyroid disease
* Diabetes mellitus
* Chronic Renal Failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-02 (Actual)

PRIMARY OUTCOMES:
visual analogue scale | 3 months
  visual analogue scale from 0-10, where 0 denoting maximum pain relief and 10 denoting no pain relief
Manchester-Oxford Foot Questionnaire | 3 months
  the Manchester-Oxford Foot Questionnaire is a 16-item instrument answered on a five-point Likert scale (each item is scored from 0 to 4, with 4 denoting 'most severe'). Scores for each item are summed to form three separate sub scales representing underlying domains: walking/standing problems (seven items), foot pain (five items), and issues related to social interaction (four items)

SECONDARY OUTCOMES:
echogenicity in longitudinal scan gray scale ultrasound | 3 months
  Hypoechogenicity was defined as a lack of the homogeneous fibrillar pattern with loss of the tightly packed echogenic lines after correcting for anisotropy. increased echogenicity is consistent with plantar fasciitis
plantar fascia thickness at the insertion in longitudinal scan of the heel | 3 months
  measurement of plantar fascia thickness at the insertion in longitudinal view of the heel. Normal thickness is ≤ 4mm. increased thickness is consistent with plantar fasciitis

CONTACTS AND LOCATIONS:
Locations (1):
- Minya university, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No